CLINICAL TRIAL: NCT00962624
Title: A Phase 2, Open-label Study of the Safety, Tolerability and Immunogenicity of a Meningococcal B Vaccine When Administered at a 0, 2, 6 Months and of a Single Dose of Meningococcal ACWY Conjugate Vaccine in Healthy Adults Aged 18-65 Years
Brief Title: Study of Meningococcal B Vaccine and ACWY Conjugate Vaccine in Healthy Adults
Acronym: MenOccy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Elizabeth Miller (Other Government)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor-Investigator, Prof. Elizabeth Miller, Prinicipal Investigator, Public Health England
Organization: Public Health England (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MenOccy; I72P1
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Meningococcal Meningitis, Serogroup A; Meningococcal Meningitis, Serogroup B; Meningococcal Meningitis, Serogroup C; Meningococcal Meningitis, Serogroup Y; Meningococcal Meningitis, Serogroup W
Keywords: Meningococcal; Vaccine; Meningitis
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis | interventions — 4CMenB vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: meningococcal B vaccine & meningococcal ACYW conjugate vaccine — Meningococcal B vaccine will be administered at 0, 2 and 6 months and a single dose of meningococcal ACYW vaccine will be administered at 0 months, concomitantly with the first dose of the meningococcal B vaccine.
  Other Names: Meningococcal ACYW vaccine- MenVeo

SUMMARY:
The study involves the measurement of immune response to vaccination with three doses of a meningococcal B vaccine and a single dose of a meningococcal ACYW conjugate vaccine in healthy adults (Laboratory workers). The study will be completed at the Manchester Medical Microbiology Partnership in the UK and will enrol staff who may be at potential occupational exposure to meningococci. Blood samples will be taken before and after each vaccination and used to determine if the vaccines induce protective responses.

DETAILED DESCRIPTION:
Laboratory staff at the Manchester Medical Microbiology Partnership may be at potential occupational exposure to meningococci. No licensed vaccine is available against serogroup B meningococci and the available plain polysaccharide serogroup ACYW vaccine is poorly immunogenic. Novartis Vaccines have developed an investigational serogroup B vaccine and a conjugated ACYW vaccine. This study will investigate these vaccines ability to induce a protective response in laboratory staff from the Manchester Medical Microbiology Partnership. Three doses of the meningococcal B vaccine will be administered at 0, 2 and 6 months and a single dose will be administered at 0 months. Blood samples will be taken before and after each vaccination and functional antibodies determined.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years of age
* Who have given written informed consent after the nature of the study has been explained.
* Who work within the Manchester Medical Microbiology Partnership and may be at potential occupational exposure to meningococci.

Exclusion Criteria:

* The possibility of pregnancy
* A serious chronic disease including progressive neurological disease or seizure disorder.
* Have a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Have a history of severe allergic reactions after previous vaccinations such as anaphylactic shock, asthma, urticaria, or other allergic reaction or hypersensitivity to any vaccine component.
* Have received another investigational agent within 90 days or before completion of the safety follow-up period in another study, whichever is longer, prior to enrollment and unwilling to refuse participation in another investigational trial through the end of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects attaining putative protective antibody concentrations against meningococci in the serum bactericidal antibody assay | one month following the last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ray Borrow, PhD, Principal Investigator — Public Health England
Locations (1):
- Manchester Medical Microbiology Partnership, Manchester, United Kingdom

REFERENCES:
- [Background] Findlow J, Bai X, Findlow H, Newton E, Kaczmarski E, Miller E, Borrow R. Safety and immunogenicity of a four-component meningococcal group B vaccine (4CMenB) and a quadrivalent meningococcal group ACWY conjugate vaccine administered concomitantly in healthy laboratory workers. Vaccine. 2015 Jun 26;33(29):3322-30. doi: 10.1016/j.vaccine.2015.05.027. Epub 2015 May 27. PMID 26025807
- [Derived] Ramirez-Bencomo F, Thistlethwaite A, Viviani V, Bartolini E, Pizza M, Biolchi A, Muzzi A, Delany I, Awanye AM, Chang CM, Borrow R, Derrick JP. Identification of immunogenic outer membrane vesicle vaccine antigen components using a meningococcal protein microarray. Vaccine. 2025 Apr 19;53:126953. doi: 10.1016/j.vaccine.2025.126953. Epub 2025 Mar 4. PMID 40043411